CLINICAL TRIAL: NCT01335035
Title: Open-Label Single-Arm Pilot Study of Deferasirox (Exjade®) in Adult Allogeneic Hematopoietic Stem Cell Transplant Recipients With Transfusional Iron Overload
Brief Title: Open-Label Single-Arm Pilot Study in Adult Allogeneic Hematopoietic Stem Cell Transplant Recipients With Transfusional Iron Overload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AES04; EudraCT: 2008-003207-30 (Registry Identifier: EudraCT)
Record Dates: First submitted 2011-03-30; First posted 2011-04-13 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Iron Overload
Keywords: Iron metabolism,; Allogenetic Hematopoietic Stem Cell Transplant,; haematological diseases
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

ARMS (1):
- ICL670 (Experimental)
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox
  Other Names: ICL670

SUMMARY:
This study has been designed to establish the efficacy and safety of deferasirox in patients with iron overload from 6 to 18 months after allogeneic hematopoietic stem cell transplant (HSCT).

The purpose of this study is to assess the mean change in serum ferritin after 52 weeks of treatment with deferasirox, in patients with iron overload (defined with serum ferritin levels ≥ 1000 ng/ml and receiving > 20 RBC concentrates) after allogeneic HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age and older
* Patients to undergo allogeneic HSCT between 6 and 18 months prior to inclusion.
* Patients with screening ANC > 1000/mm3 and ferritin values ≥ 1000 ng/mL (ferritin values must be measured in two measurements at one-week intervals).
* Patients receiving at least 20 RBC concentrate units or 100mL/kg RBC during their lives.
* Patients giving their informed consent (prior to performing any study procedure)

Exclusion Criteria:

* Haemosiderosis not related to transfusion.
* Patients with concomitant active malignancy.
* Active known viral hepatitis or known HIV-positive.
* Mean levels of alanine aminotransferase (ALT) > 5x ULN
* Treatment with any iron chelating agent after allogeneic HSCT.
* Uncontrolled hypertension.

Other protocol-defined inclusion/exclusion criteria may app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean change in serum ferritin | after 52 weeks of treatment with deferasirox

SECONDARY OUTCOMES:
Mean change in the no. of sideroblasts, assessed by Perls staining | after 52 weeks of treatment with deferasirox
Mean change in liver iron concentration (LIC), assessed by liver MRI. | after 52 weeks of treatment with deferasirox
Incidence of chronic graft-versus-host disease ("limited" or "extensive", according to Shulman criteria) | up to 52 weeks of study
Incidence of infections (bacterial, viral, or fungal) | up to 52 weeks of study
Incidence of venous occlusive disease during the study | up to 52 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Spain (9):
  - Novartis Investigative Site, Andalucia
  - Novartis Investigative Site, Asturias
  - Novartis Investigative Site, Canarias
  - Novartis Investigative Site, Castilla Y Leon
  - Novartis Investigative Site, Cataluna
  - Novartis Investigative Site, Comunidad Valenciana
  - Novartis Investigative Site, Islas Baleares
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia

REFERENCES:
- [Derived] Vallejo C, Batlle M, Vazquez L, Solano C, Sampol A, Duarte R, Hernandez D, Lopez J, Rovira M, Jimenez S, Valcarcel D, Belloch V, Jimenez M, Jarque I; Subcommittee of Non-Infectious Complications of the Grupo Espanol de Trasplante Hematopoyetico (GETH). Phase IV open-label study of the efficacy and safety of deferasirox after allogeneic stem cell transplantation. Haematologica. 2014 Oct;99(10):1632-7. doi: 10.3324/haematol.2014.105908. Epub 2014 Jul 4. PMID 24997153